CLINICAL TRIAL: NCT06577246
Title: Effects of Periodontal Disease Prediction System on Oral Hygiene Motivation in Patients With Periodontitis: A Prospective Randomised Controlled Clinical Study
Brief Title: Assessment of the Effect of Periodontal Disease Prediction System on Oral Hygiene Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Abant Izzet Baysal University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Şadiye GÜNPINAR, principal ınvestigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGUNPINAR/119S025
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Motivational Interviewing; Computer-Aided Design; Periodontal Diseases
Keywords: Oral hygiene motivation; computer-aided design; periodontal disease; motivational interview
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Method (CM) (Active Comparator): Individuals in this group receive instructions on oral care after initial periodontal treatment from the physician (SG) who is familiar with the patient groups. The physician verbally explains the development of periodontal disease, its causes, symptoms, and the potential consequences of irregular oral care, using a brochure to reinforce these points.
  Interventions: Procedure: scaling root planing
- Three-Dimensional Animation (3DA) (Active Comparator): The video used in the study was created by DentalMaster (MD Stimulation Ltd) by combining their own footage (http://www.mdsimulation.com/). This video is divided into three parts, summarized below:
  * i. Overview of the causes and symptoms of periodontal disease (section 1)
  * ii. Treatment of periodontal disease and daily oral care practices for individuals (section 2)
  * iii.Consequences of periodontal disease (such as gingival recession and tooth loss) that individuals may face if periodontal diseases are not treated and if they do not perform regular oral care (section 3). In this group, patients watch the video together with the physician (SG), who is familiar with the randomized patient groups.
  Interventions: Procedure: scaling root planing; Behavioral: Three-Dimensional Animation (video1-2); Behavioral: Three-Dimensional Animation (video 3)
- Periodontal Disease Prediction (PDP) (Experimental): The patients in the test group viewed sections 1 and 2 videos in the same manner as the 3DA group. However, unlike the 3DA group, they did not view section 3. Instead, they were shown estimates of their current condition and potential future periodontal tissue loss (gingival recession) for 1-5 years, 5-10 years, and 10-20 years (1). These projections were presented to the patients in three dimensions with PDP visualisation.
  Interventions: Procedure: scaling root planing; Behavioral: Three-Dimensional Animation (video1-2); Behavioral: Periodontal Disease Prediction (PDP)

INTERVENTIONS:
Procedure: scaling root planing — periodontal treatment in all groups was performed using ultrasonic and hand instruments (#15/30, #6/7) by the same physician (UGE) who was blind to the study groups.
Behavioral: Three-Dimensional Animation (video1-2) — The video used in the study was created by DentalMaster (MD Stimulation Ltd) by combining their own footage (http://www.mdsimulation.com/). This video is divided into three parts, summarized below:
  * i. Overview of the causes and symptoms of periodontal disease (section 1)
  * ii. Treatment of periodontal disease and daily oral care practices for individuals (section 2)
  Arms: Periodontal Disease Prediction (PDP); Three-Dimensional Animation (3DA)
Behavioral: Three-Dimensional Animation (video 3) — iii.Consequences of periodontal disease (such as gingival recession and tooth loss) that individuals may face if periodontal diseases are not treated and if they do not perform regular oral care (section 3). In this group, patients watch the video together with the physician (SG), who is familiar with the randomized patient groups.
  Arms: Three-Dimensional Animation (3DA)
Behavioral: Periodontal Disease Prediction (PDP) — The patients in the test group viewed sections 1 and 2 videos in the same manner as the 3DA group. However, unlike the 3DA group, they did not view section 3. Instead, they were shown estimates of their current condition and potential future periodontal tissue loss (gingival recession) for 1-5 years, 5-10 years, and 10-20 years. These projections were presented to the patients in three dimensions with PDP visualisation.
  Arms: Periodontal Disease Prediction (PDP)

SUMMARY:
The aim of this trial is to evaluate the effect of patient specific periodontal disease prediction (PDP) system, a part of motivational interview, (MI) on probing depth (PD), Rustogi modified Navy Plaque Index (RMNPI), and papillary bleeding index (PBI) scores in patients with periodontitis following non-surgical periodontal therapy.

DETAILED DESCRIPTION:
A total of 120 participants included in our study and were then randomly assigned to three groups: a) conventional method (CM) (n=40), b) three-dimensional animation (3DA) (n=40), and c) Periodontal Disease Prediction (PDP) interaction (n=40). PD, PBI, and RMNPI values were recorded before periodontal therapy (T0). Following periodontal treatment, individuals in the CM group were instructed on oral hygiene via a model and brochure. Individuals in the 3DA group were informed using 3D video visuals. Participants in the PDP group were informed in a computer-based three-dimensional manner, providing projections of their current status and potential future gingival recessions after viewing the first and second parts of the 3D animation. Clinical periodontal measurements were repeated at 3, 6, and 12 months post-treatment. Data obtained after the study were analyzed using appropriate statistical methods. It was concluded that the proposed approach in this project could enhance periodontitis individuals' awareness about periodontal disease and personal oral hygiene especially for interdental cleaning over a long period. By this way, this PDP system can lead clinical benefits in reducing the recurrence of periodontal disease. It was hypothesized that patients in the PDP group could achieve significantly better plaque control and have lower bleeding scores compared to patients in the control groups, which include traditional oral hygiene motivation and three-dimensional video education.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 to 60 years.
* No prior periodontal treatment or oral hygiene education.
* Simplified Oral Hygiene Index (OHI-S) greater than 3 (indicating poor oral hygiene).
* Diagnosed with 'Stage III' 'Grade B' periodontitis.
* At least 20 natural teeth present (excluding third molars).
* Minimum of 12 years of education.
* Not a dentist or dental student.
* No systemic diseases affecting memory or cognitive function.
* No physical disabilities that could hinder the performance of oral hygiene procedures.

Exclusion Criteria:

* Presence of diffuse dentinal hypersensitivity.
* Acute infections.
* Faulty restorations.
* Root caries complicating oral hygiene.
* Full-mouth fixed or removable dentures.
* Ongoing orthodontic treatment.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
rustogi modified navy plaque index (RMNPI) | baseline (T0) and repeated at 3rd (T1), 6th (T2) and 12th (T3) months
  RMNPI was assessed using a specialized plaque staining agent on each of the nine sites on both buccal and lingual tooth surfaces. The individual mean PI was calculated by scoring the presence of plaque at each site as '1' and its absence as '0', then dividing by the total number of surfaces evaluated. Using this index, PI can be separately calculated for the entire mouth (A-I), the gingival margin (A-C), interproximal areas (D and F), and surfaces that come into contact with dental floss (A, C, D, and F)

SECONDARY OUTCOMES:
Probing depth (PD) | baseline (T0) and repeated at 3rd (T1), 6th (T2) and 12th (T3) months
  PD measurements was evaluated at six regions of each tooth
bleeding on probing (BoP) | baseline (T0) and repeated at 3rd (T1), 6th (T2) and 12th (T3) months
  BoP associated with PD measurements was evaluated at six regions of each tooth as presence/absence and recorded as %.
papillary bleeding index (PBI) | baseline (T0) and repeated at 3rd (T1), 6th (T2) and 12th (T3) months
  PBI is calculated by scoring the papillae in the facial/buccal and palatinal/lingual regions of each tooth based on the presence or absence of bleeding from probing and the overall condition of the gingiva. The average PBI value for an individual was calculated by dividing the total sum of the values by the number of papillae assessed.
Gingival ındex (GI) | baseline (T0) and repeated at 3rd (T1), 6th (T2) and 12th (T3) months
  Each tooth's mesial, distal, buccal, and lingual gingival margins are evaluated. These values are then summed and divided by four. This process calculates the Gingival Index (GI) for each tooth. When the total of these values is divided by the number of teeth, the individual's GI score is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Asc. Prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Gunpinar S, Sevinc AS, Akgul Z, Tasmektepligil AA, Gunpinar E. Patient-specific gingival recession system based on periodontal disease prediction. Int J Comput Dent. 2025 Apr 3;28(1):35-45. doi: 10.3290/j.ijcd.b4784721. PMID 38112604